CLINICAL TRIAL: NCT06780748
Title: Photo-medicine-Guided Dual Approach for Reoperation of Sentinel Lymph Nodes in Locally Recurrent Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Seeyoun Lee, Doctor, M.D., head of center for breast cancer, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC-2310621-2
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer; Locally Recurrent Breast Cancer; Sentinel Lymph Node Biopsy (SLNB); Reoperation; ICG (indocyanine Green)
Keywords: Breast cancer; Locally Recurrent Breast cancer; Sentinel Lymph Node Biopsy (SLNB); Reoperation; ICG(indocyanine green)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radioactive Isotope (RI) with Indocyanine Green Fluorescence (ICG-F) (Experimental): Sentinel lymph node mapping using a combination of radioactive isotope and indocyanine green fluorescence (ICG-F)
  Interventions: Procedure: Identification rate of sentinel lymph node

INTERVENTIONS:
Procedure: Identification rate of sentinel lymph node — To evaluate the identification rate of sentinel lymph nodes (SLNs). The study will compare the identification rates based on different localization techniques for SLN mapping

SUMMARY:
Sentinel lymph node biopsy (SLNB) is essential for staging and treatment planning in early breast cancer patients. As a less invasive procedure, it has replaced axillary lymph node dissection (ALND) by reducing complications and improving patient outcomes. However, the 10-year local recurrence rate for breast cancer is approximately 2-10%, and the role of SLNB in the surgical management of recurrent breast cancer remains unclear.

According to the NCCN guidelines and Korean Breast Cancer Treatment Recommendations, surgical management for recurrent breast cancer includes mastectomy and axillary lymph node surgery for patients who have previously undergone breast-conserving surgery and radiotherapy. For axillary recurrence, surgery is recommended if feasible, followed by radiotherapy. Conversely, the ASCO guidelines recommend SLNB for surgically resectable recurrent breast cancer, and recent studies have reported promising outcomes for repeat sentinel lymph node biopsy (reSLNB). Vugts G et al. demonstrated an 80.1% tumor-negative rate with reSLNB, suggesting that ALND could be avoided in many cases.

Although reSLNB offers the advantage of reducing unnecessary invasive procedures and associated complications, challenges remain due to disrupted lymphatic pathways in patients who have previously undergone surgery and radiotherapy. Additionally, research on the long-term prognosis of these patients is still limited.

This study aims to evaluate the detection rate of sentinel lymph nodes using a photo-medicine-based dual localization technique that combines traditional radiotracer methods with indocyanine green-fluorescence (ICG-F) in patients undergoing reSLNB for locally recurrent breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ipsilateral locally recurrent breast cancer who previously underwent ipsilateral axillary surgery.
* Female patients aged 18 years or older.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients who voluntarily decide to participate in the study and provide written informed consent.

Exclusion Criteria:

* Patients with distant metastases.
* Patients who previously underwent ipsilateral mastectomy.
* Pregnant or breastfeeding women.
* Patients with a general condition that impairs the ability to understand or provide informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification Rate of Sentinel Lymph Nodes (SLNs) | Day of Surgery

SECONDARY OUTCOMES:
Comparison of Identification Rates Based on Sentinel Lymph Node Localization Techniques | Day of Surgery

CONTACTS AND LOCATIONS:
Overall Officials: SEEYOUN LEE, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided